CLINICAL TRIAL: NCT01132911
Title: A Phase I Study of Vorinostat and Bortezomib in Children With Refractory of Recurrent Solid Tumors, Including CNS Tumors and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100119; 10-C-0119
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-13

CONDITIONS: Lymphoma; Sarcoma; WilmsTumor; Neuroblastoma
Keywords: Solid Tumors; Maximum Tolerated Dose; Lymphoma; Dose Escalation; Pharmacokinetics; Pediatric Cancer; Solid Tumor; Sarcoma; Wilms Tumor; Neuroblastoma
MeSH Terms: conditions — Lymphoma; Sarcoma; Neuroblastoma; Neoplasms; Wilms Tumor | interventions — Vorinostat; Bortezomib

INTERVENTIONS:
Drug: Vorinostat (SAHA)
Drug: Velcade (PS-341, Bortezomib)

SUMMARY:
Background:

- Vorinostat and bortezomib are anti-tumor drugs that have been approved by the Food and Drug Administration to treat different kinds of myeloma and lymphoma in adults. The combination of these two drugs has been tried in a small number of adults, but it has not been formally approved and is experimental, particularly in children. Researchers are interested in determining safe and effective treatment doses of vorinostat and bortezomib in children, and learning more about how these drugs affect tumor growth and human development.

Objectives:

* To determine safe and effective doses of vorinostat and bortezomib to treat solid tumors in children.
* To study the effects of vorinostat and bortezomib on blood cells, blood flow, and human development.

Eligibility:

- Children, adolescents, and young adults between 1 and 21 years of age who have been diagnosed with solid tumors that have not responded to treatment.

Design:

* Eligible participants will be screened with a physical examination, blood and tumor samples, and imaging studies.
* Participants will have 21-day treatment cycles of vorinostat and bortezomib. Vorinostat will be given as either tablets or liquid doses on days 1 through 5 and 8 through 12 of each cycle. Bortezomib will be given as an intravenous injection on days 1, 4, 8, and 11 of each cycle. Participants will keep a drug administration diary to record information about side effects or other problems with the treatment.
* Participants may continue to receive vorinostat and bortezomib for up to 2 years unless serious side effects develop or the tumor does not respond to treatment.
* Additional blood samples will be taken at regular intervals for the first 3 days after the first bortezomib dose and for the first 2 days after the first vorinostat dose of the first treatment cycle.

DETAILED DESCRIPTION:
Background:

-The combination of vorinostat and bortezomib has been shown to be synergistic in vitro in a variety of malignancies, including hepatoma, multiple myeloma, leukemia, lymphoma, and gastrointestinal cancer. Currently several phase 2 adult studies are underway evaluating combination therapy.

Objectives:

* To determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose of the combination of oral vorinostat administered on days 1-5 and 8-12 and bortezomib administered intravenously on days 1, 4, 8, 11, every 21 days to children with refractory or recurrent solid tumors.
* To define and describe the toxicities of vorinostat in combination with bortezomib administered on this schedule.
* To characterize the pharmacokinetics of vorinostat and bortezomib in combination in children with refractory or recurrent solid tumors.
* Secondary objectives include preliminary definition of the antitumor activity of these agents when administered together; and assessment of the biologic activity of bortezomib by measuring NF-kappaB activity in peripheral blood mononuclear cells (PBMC) and by measuring endoplasmic reticulum stress response using the GRP78 molecular chaperone marker in PBMC.

Eligibility:

* Patients greater than12 months and less than or equal to 21 years of age with a diagnosis and histologic verification (except patients with instrinsic brain stem tumors, optic pathway gliomas or pineal tumors) of measureable or evaluable relapsed or refractory solid tumors including CNS tumors and lymphomas are eligible. Current disease state must be one for which there is no known curative therapy, or therapy proven to prolong survival.
* Performance score: Karnofsky greater than or equal to 60% for patients greater than 16 years of age; Lansky greater than or equal to 60 for patients less than or equal to 16 years of age.
* Must have fully recovered from acute toxic effects from all prior therapy which have been completed within the specified prior time frame. Have adequate organ function as determined by laboratory evaluation.

Design:

* This is a phase I study of vorinostat administered orally once daily on days 1-5 and day 8-12 in combination with bortezomib administered intravenously on days 1, 4, 8, and 11 of a 21 day cycle. Disease evaluation will be performed after cycle 1 and then every 2 cycles thereafter.
* Therapy may continue for up to 2 years in the absence of progressive disease or unacceptable toxicity.
* Optional participation in correlative biology studies or pharmacokinetic studies will be offered.

ELIGIBILITY:
* Eligibility Criteria:

Inclusion Criteria:

* Patients older than12 months and less than or equal to 21 years of age with a diagnosis and histologic verification (except patients with instrinsic brain stem tumors, optic pathway gliomas or pineal tumors) of measureable or evaluable relapsed or refractory solid tumors including CNS tumors and lymphomas are eligible.
* Current disease state must be one for which there is no known curative therapy, or therapy proven to prolong survival.
* Performance score: Karnofsky greater than or equal to 60% for patients greater than 16 years of age; Lansky greater than or equal to 60 for patients less than or equal to 16 years of age.
* Must have fully recovered from acute toxic effects from all prior therapy which have been completed within the specified prior time frame.
* Have adequate organ function as determined by laboratory evaluation.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2010-05-10; Primary Completion 2011-04-13 (Actual); Study Completion 2011-04-13 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose and Phase 2 dose of combination vorinostat and bortezomib to children with refractory or recurrent solid tumors.
Define toxicities and pharmacokinetics.

SECONDARY OUTCOMES:
To define antitumor activity, assess biological activity of bortezomib by measuring NF-kb activity in PBMC and to assess the biologic activity of bortezomib by measuring endoplasmic reticulum stress response using GRP78 molecular chaperone marke...

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Emanuele S, Lauricella M, Carlisi D, Vassallo B, D'Anneo A, Di Fazio P, Vento R, Tesoriere G. SAHA induces apoptosis in hepatoma cells and synergistically interacts with the proteasome inhibitor Bortezomib. Apoptosis. 2007 Jul;12(7):1327-38. doi: 10.1007/s10495-007-0063-y. PMID 17351739
- [Background] Pei XY, Dai Y, Grant S. Synergistic induction of oxidative injury and apoptosis in human multiple myeloma cells by the proteasome inhibitor bortezomib and histone deacetylase inhibitors. Clin Cancer Res. 2004 Jun 1;10(11):3839-52. doi: 10.1158/1078-0432.CCR-03-0561. PMID 15173093
- [Background] Mitsiades CS, Mitsiades NS, McMullan CJ, Poulaki V, Shringarpure R, Hideshima T, Akiyama M, Chauhan D, Munshi N, Gu X, Bailey C, Joseph M, Libermann TA, Richon VM, Marks PA, Anderson KC. Transcriptional signature of histone deacetylase inhibition in multiple myeloma: biological and clinical implications. Proc Natl Acad Sci U S A. 2004 Jan 13;101(2):540-5. doi: 10.1073/pnas.2536759100. Epub 2003 Dec 26. PMID 14695887